CLINICAL TRIAL: NCT06752096
Title: Robot-assisted Neurovascular Intervention for Patients Indicated for Angiography, Cerebral Artery Embolization, and Thrombectomy: Exploratory Study to Compare to Existing Interventional Procedures
Brief Title: Robot-Assisted Neurovascular Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Navigantis Inc. (Industry)
Collaborators: Severance Hospital, Yonsie University College of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024-2751-002
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Meningioma; Neurovascular Disorder
Keywords: Robot-assisted neurovascular Intervention; cerebral angiogram; Meningioma; Thrombectomy; Ischemic Stroke
MeSH Terms: conditions — Stroke; Meningioma; Ischemic Stroke | interventions — Cerebral Angiography; Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (1):
- Robot Assisted Neurovascular Intervention (Experimental): Patients will undergo robot-assisted neurovascular interventions.
  Interventions: Procedure: cerebral angiography, arterial embolization, thrombectomy; Device: Cerebral angiogram using robotic device; Device: Meningioma embolization using robotic device.; Device: Mechanical thrombectomy for stroke using a robotic device.

INTERVENTIONS:
Procedure: cerebral angiography, arterial embolization, thrombectomy — This intervention will be conducted using robotic navigation.
Device: Cerebral angiogram using robotic device — Diagnostic cerebral angiogram will be performed using a robot to navigate guidewires and catheters to target vessels.
Device: Meningioma embolization using robotic device. — Meningioma tumors will be embolized using a robot to navigate catheters and wires to the target vessels to the tumor.
Device: Mechanical thrombectomy for stroke using a robotic device. — Mechanical thrombectomy procedure will use a robot to navigate catheters, guidewires, and thrombectomy devices to the target vessel.

SUMMARY:
Patients scheduled for neurovascular interventions may be eligible to have their procedure done robotically.

DETAILED DESCRIPTION:
Patients scheduled for manual neurovascular interventions, such as diagnostic cerebral angiography for cerebrovascular diseases, arterial embolization for meningioma treatment, and thrombectomy for thrombotic arterial occlusion-induced cerebral ischemia, may be considered to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for neurovascular interventions, such as diagnostic cerebral angiography for cerebrovascular diseases, arterial embolization for meningioma treatment, and thrombectomy for thrombotic arterial occlusion-induced cerebral ischemia, are selected according to the same criteria as standard cerebral angiography and interventional procedures.

Exclusion Criteria:

Exclusion Criteria 1 (General):

1. Patients who have undergone surgery within 4 weeks prior to study participation or have not fully recovered from surgery.
2. Patients who are pregnant or breastfeeding.
3. Patients with existing or anticipated vasospasm, bleeding, or severe atheromatous disease.
4. Patients allergic to contrast agents used in angiography.
5. Patients with renal failure.
6. Patients with a history of cardiac events, such as myocardial infarction or superior vena cava (SVC) syndrome, within 3 months prior to study participation, or with existing heart disease.
7. Patients unable to cooperate due to difficulty in expressing intent to the extent that the procedure cannot proceed.
8. Patients with severe or life-threatening comorbidities that could significantly affect symptom improvement or render the procedure unbeneficial.
9. Patients with non-life-threatening comorbidities that prevent proper follow-up for treatment.

Exclusion Criteria 2 (Cerebral Ischemic Stroke Patient):

1. Patients with an ASPECTS score of 0-2 on a pre-treatment non-contrast CT.
2. Inability to perform femoral puncture within 60 minutes of completing CT angiography (if CT perfusion is performed, it must be done after CT angiography).
3. Absence of a femoral pulse.
4. Cases where vascular access is highly challenging, with an anticipated time exceeding 90 minutes from CT angiography to reperfusion.
5. Patients suspected to have cerebral artery dissection or atherosclerosis as the cause of stroke.
6. Patients where the intracranial occlusion is determined to be chronic based on clinical history, prior imaging, or clinical judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Success rate of target vessel access | From enrollment through end of procedure.
  Measurement Parameters: The primary outcome assesses whether the Vasco Robotic system navigates catheter or other procedural devices successfully to the target vessel.

CONTACTS AND LOCATIONS:
Locations (1):
- Severence Hospital, Yonsei University College of Medicine, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: Undecided